CLINICAL TRIAL: NCT04921423
Title: To Investigate the Effect of Situational Simulation Teaching Intervention on Nursing Students' Attitude and Empathy Towards the Elderly
Brief Title: The Study on the Attitude and Empathy of Nursing Students Towards the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chia Jung Hsieh, PhD, RN, Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SMHIRB109012
Record Dates: First submitted 2021-05-20; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Empathy; Attitude
Keywords: situational simulation teaching; Attitude towards the elderly; Empathy towards the elderly
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- situational simulation teaching (Experimental): Clinical case role play and empathy skill practice
  Interventions: Behavioral: Situational simulation teaching
- Clinical Case (Problem Based Learning) (No Intervention): Clinical Case discuss (Problem Based Learning)

INTERVENTIONS:
Behavioral: Situational simulation teaching — The intervention included communication theory and skills, aging trend and knowledge, teaching plans for elderly nursing, activities for the elderly and visual experience, application and debriefing of empathy.
  Arms: situational simulation teaching

SUMMARY:
The effect of situational simulation teaching intervention on the attitude and empathy of nursing students towards the elderly can be divided into two stages. The first stage is a cross-sectional study on the aging knowledge, attitude and empathy of nursing students. The second stage was the change of nursing students' attitude and empathy towards the elderly after the intervention of situational simulation teaching. The intervention measures included communication theory and skills, aging trend and knowledge, teaching plans for elderly nursing, activities for the elderly and visual experience, application and debriefing of empathy. This study collected and analyzed the data of aging knowledge, attitude and empathy towards the elderly at the end of the term and one month later, in order to explore the changes of attitude and empathy towards the elderly of nursing students after the intervention of situational simulation teaching.

DETAILED DESCRIPTION:
Taiwan has entered an aging society and will enter a super aging society in 2026. With the increase of chronic diseases and aging of the elderly, they are gradually weakened. When they are unable to take care of themselves in the future, the demand for institutional care is increasing, and the future labor force is gradually decreasing. The training of care manpower is facing a test. The purpose of this study is to explore the aging knowledge, attitude towards the elderly and empathy of nursing students, and then to explore the change of students' aging knowledge, attitude towards the elderly and empathy after the intervention of simulated situational teaching course, and to explore the change of their willingness to join the elderly career in the future.

In the first stage, a cross-sectional study was conducted to extract 139 nursing science students from an Eastern college. In order to explore the aging knowledge, attitude and empathy towards the elderly, and future career involvement willingness of nursing students, Pearson product difference correlation analysis and Spearman grade correlation coefficient analysis were used to predict the relationship between variables, and multiple linear regression model was used to analyze the data. In the second stage of the study, the subjects were the same as those in the first stage. The experimental group and the control group were randomly assigned by drawing lots, with at least 51 participants. At the beginning, the end and one month after the course, we explored the change of students' ability to take care of the elderly and their willingness to devote to the elderly related career in the future. For inferential analysis, independent sample t-test and chi square test were used to analyze whether there were statistically significant differences in basic information, aging knowledge and attitude towards the elderly between the intervention group and the control group, and then generalized estimating equation (GEE) was used to check the effectiveness of situational simulation course after controlling relevant interference factors. It is expected that nursing students can experience the inconvenience of daily life of the elderly in the way of situational simulation, use empathy skills, carry out role play of teaching plan, and simulate the care behavior and empathy of the elderly in the clinical situation, so as to improve their willingness to choose jobs related to the elderly after graduation.

ELIGIBILITY:
Inclusion Criteria:

* Sophomores of Nursing College

Exclusion Criteria:

* Students with nursing practice experience

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 142 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-04-04 (Actual); Study Completion 2021-06-25 (Estimated)

PRIMARY OUTCOMES:
The Aging knowledge | baseline, pre-intervention(T0)
  The Aging Knowledge Questionnaire contains 16 true or false questions, and each correct answer gets one point. The higher the score, the better the knowledge of aging. There is no subscale. The score of range from 0-16.
The Aging knowledge | through study completion, an average of 4 months(T1)
  The Aging Knowledge Questionnaire contains 16 true or false questions, and each correct answer gets one point. The higher the score, the better the knowledge of aging. There is no subscale. The score of range from 0-16.
The Aging knowledge | One month after the completion of the intervention(T2)
  The Aging Knowledge Questionnaire contains 16 true or false questions, and each correct answer gets one point. The higher the score, the better the knowledge of aging. There is no subscale. The score of range from 0-16.
Old People Scale | baseline, pre-intervention(T0)
  There are 11 questions in the scale of attitude towards the elderly. The higher the score of Likerts Scale 1-7, the more negative the attitude towards the elderly. The score of range from 1-49.
Old People Scale | through study completion, an average of 4 months(T1)
  There are 11 questions in the scale of attitude towards the elderly. The higher the score of Likerts Scale 1-7, the more negative the attitude towards the elderly.The score of range from 1-49.
Old People Scale | One month after the completion of the intervention(T2)
  There are 11 questions in the scale of attitude towards the elderly. The higher the score of Likerts Scale 1-7, the more negative the attitude towards the elderly.The score of range from 1-49.
Chinese Version of the Jefferson Scale of Empathy | baseline, pre-intervention(T0)
  There are 20 questions in the empathy scale consists of three sub-scales.The higher the score of Likerts Scale 1-7, the better the empathy. The score of range from 1-140.
Chinese Version of the Jefferson Scale of Empathy | through study completion, an average of 4 months(T1)
  There are 20 questions in the empathy scale consists of three sub-scales.The higher the score of Likerts Scale 1-7, the better the empathy.The score of range from 1-140.
Chinese Version of the Jefferson Scale of Empathy | One month after the completion of the intervention(T2)
  There are 20 questions in the empathy scale consists of three sub-scales.The higher the score of Likerts Scale 1-7, the better the empathy.The score of range from 1-140.

SECONDARY OUTCOMES:
Clinical Situational Empathy Scales | One month after the completion of the intervention(T2)
  There are two teaching plans of the Clinical Situation Empathy Scale, which has 4 subs-cales and total of 32 questions. The score of the Likerts Scale is 1-4, and the higher the score, the better the demonstration of empathy.The score of range from 1-128.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Jung Hsieh, PhD, Study Director — National Taipei University of Nursing and Health Sciences
Locations (1):
- St. Mary's Medicine Nursing and Management College, Yilan, Sanxing Township, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeffries PR. A framework for designing, implementing, and evaluating simulations used as teaching strategies in nursing. Nurs Educ Perspect. 2005 Mar-Apr;26(2):96-103. PMID 15921126
- [Background] Cant RP, Cooper SJ. Simulation-based learning in nurse education: systematic review. J Adv Nurs. 2010 Jan;66(1):3-15. doi: 10.1111/j.1365-2648.2009.05240.x. PMID 20423432
- [Background] Lee KC, Yu CC, Hsieh PL, Li CC, Chao YC. Situated teaching improves empathy learning of the students in a BSN program: A quasi-experimental study. Nurse Educ Today. 2018 May;64:138-143. doi: 10.1016/j.nedt.2018.02.013. Epub 2018 Feb 13. PMID 29476960
- [Background] Zhang S, Liu YH, Zhang HF, Meng LN, Liu PX. Determinants of undergraduate nursing students' care willingness towards the elderly in China: Attitudes, gratitude and knowledge. Nurse Educ Today. 2016 Aug;43:28-33. doi: 10.1016/j.nedt.2016.04.021. Epub 2016 May 2. PMID 27286941
- [Background] Mennenga HA, Bassett S, Pasquariello L. Empathy Development Through Case Study and Simulation. Nurse Educ. 2016 May-Jun;41(3):139-42. doi: 10.1097/NNE.0000000000000226. PMID 26448156
- [Background] Elliott R, Bohart AC, Watson JC, Greenberg LS. Empathy. Psychotherapy (Chic). 2011 Mar;48(1):43-9. doi: 10.1037/a0022187. PMID 21401273